CLINICAL TRIAL: NCT06256497
Title: Revita DMR Post Market Pilot Clinical Registry
Brief Title: A Prospective Study to Evaluate Revita DMR Post Market Pilot Clinical Follow-Up Registry in Patient With Type 2 Diabetes
Status: Suspended | Type: Observational
Why Stopped: The company paused enrollment due to a strategic decision to pause commercialization in the EU and specifically Germany. The company will follow currently enrolled subjects per protocol.
Sponsor: Fractyl Health Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: C-00075
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 Diabetes; DMR; Duodenal Mucosal Resurfacing; Revita
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- DMR Treated Patients
  Interventions: Device: Duodenal Mucosal Resurfacing (DMR)

INTERVENTIONS:
Device: Duodenal Mucosal Resurfacing (DMR) — The Revita System is a hydrothermal ablation system, (CE) certified, intended to impart insulin-sensitizing properties to the body via ablation & rejuvenation of the duodenal mucosa. As an adjunct to diet and exercise, Revita is intended to 1. improve glycemic control in patients with T2D who have preserved pancreatic beta cell function and whose diabetes is inadequately controlled despite oral and/or injectable glucose lowering medications and/or long-acting insulin therapy, 2. Reduce liver fat in patients with T2D and Non-Alcoholic Fatty Liver Disease (NAFLD). The single use Revita Catheter and Line Set are provided sterile and are not implantable or reusable. These disposables are used with the Revita Console an electromechanical device that controls the ablation cycle and submucosal expansion. The Revita System is used in a suitably equipped endoscopy suite. The Catheter contacts the patient's digestive tract for approximately 45-60 minutes.
  Other Names: Revita DMR

SUMMARY:
The Revita DMR Post Market Pilot Clinical Registry is a post-market, prospective, observational, noninterventional clinical registry in patients with T2D in Germany undergoing the Revita Procedure with the CE marked Revita System (Fractyl Health, Lexington, MA, USA) in accordance with its intended purposes. Patient's participation in this study has no impact on his or her indication or opportunity to receive therapy. Patients are to be treated in compliance with the current Revita System's IFU of the CE marked Revita System as well as according to medical society guidelines and physician discretion.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent in accordance with GCP and local legislation
* Adults (≥18 years) with the diagnosis of T2D
* BMI of <=45 kg/m2 at the time of presentation/screening
* T2D mellitus inadequately controlled on therapy (HbA1c ≥7.0 and ≤10.0% [53-86 mmol/mol] at the time of initial presentation for screening and with the need for therapy escalation [dose increase of existing therapy or additional prescription of insulin and/or OADs or change of therapy regimen]) to achieve the therapeutic HbA1c target defined by the physician
* Treatment with oral and/or injectable glucose lowering medications and/or long-acting insulin therapy

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with T2D in Germany undergoing the Revita Procedure with the CE marked Revita System (Fractyl Health, Lexington, MA, USA) in accordance with its intended purposes and meeting the study inclusion and exclusion criteria below. Patient's participation in this study has no impact on his or her indication or opportunity to receive therapy. Patients are to be treated in compliance with the current Revita System's IFU of the CE marked Revita System as well as according to medical society guidelines and physician discretion.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Clinical effectiveness | Baseline, 1, 3-, 6-, 12-, and 24-months post-procedure.
  Improvement in glycemic control measured by fasting blood glucose (FPG)
Clinical effectiveness | Baseline, 1, 3-, 6-, 12-, and 24-months post-procedure.
  Improvement in glycemic control measured by HbA1c, random glucose (non-fasting),
Clinical effectiveness | Baseline, 1, 3-, 6-, 12-, and 24-months post-procedure.
  Improvement in glycemic control measured by fasting insulin
Clinical effectiveness | Baseline, 1, 3-, 6-, 12-, and 24-months post-procedure.
  Improvement in glycemic control measured by fasting plasma glucagon
Clinical effectiveness | Baseline, 1, 3-, 6-, 12-, and 24-months post-procedure.
  Improvement in glycemic control measured by C-peptide.
Clinical effectiveness | Baseline, 1, 3-, 6-, 12-, and 24-months post-procedure.
  Changes in antidiabetic medication dosages

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Martin, MD, Principal Investigator — Head of Diabetology and Director of the West-German Diabetology and Health Center (WDGZ); Jochen Seufert, MD, Study Chair — Department Head Endocrinology and Diabetology, University Hospital Freiburg
Locations (1):
- Westdeutsches Diabetes und Gesundheitszentrum, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No